CLINICAL TRIAL: NCT05962957
Title: Clinical Study to Compare the Possible Safety and Efficacy of Pentoxifylline and Celecoxib in Patients With Parkinson's Disease Treated With Conventional Treatment
Brief Title: Role of Pentoxifylline and Celecoxib in Parkinsonism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Collaborators: Tanta University (Other); Mohanad Omar Khrieba Clinical Pharmacy Department, Faculty of Pharmacy - Horus University (Unknown)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Teaching assisstant, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1235
Record Dates: First submitted 2023-07-16; First posted 2023-07-27 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; Pentoxifylline; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): control group ( levo-dopa group, n =25 ) who will receive levo-dopa/carbidopa (125/12.5) mg three times daily for 6 months.
  Interventions: Drug: carbidopa-levodopa
- PTX group (Active Comparator): (Pentoxyifylline group, n= 25) will receive levo-dopa/carbidopa (125/12.5) mg three times daily plus pentoxifylline 400 mg two times daily for 6 months.
  Interventions: Drug: carbidopa-levodopa; Drug: Pentoxifylline 400 MG
- Celecoxib group (Active Comparator): will receive levo-dopa/carbidopa (125/12.5) mg three times daily plus celecoxib 200 mg once daily for 6 months.
  Interventions: Drug: carbidopa-levodopa; Drug: Celecoxib 200mg

INTERVENTIONS:
Drug: carbidopa-levodopa — Levodopa is typically prescribed to a patient with Parkinson disease once symptoms become more difficult to control with other anti-parkinsonism drugs. The drug can also be used for postencephalitic parkinsonism and symptomatic parkinsonism due to carbon monoxide intoxication
Drug: Pentoxifylline 400 MG — Pentoxifylline (PTX) has a well validated immune modulatory and anti-inflammatory efficacy via suppression of the TLR4/NF-κB network signaling pathway. Moreover, Pentoxifylline has a potential antioxidant capacity mostly via nuclear erythroid 2-related factor 2 (Nrf2) activation with subsequent up-regulation and expression of several antioxidant enzymes
  Arms: PTX group
Drug: Celecoxib 200mg — Celecoxib is a nonsteroidal anti-inflammatory drug (NSAID) used to treat mild to moderate pain and help relieve symptoms of arthritis
  Arms: Celecoxib group

SUMMARY:
Parkinson's disease (PD) is a chronic neurodegenerative disease clinically characterized by bradykinesia, hypokinesia, rigidity, resting tremor, and postural instability. These motor manifestations are attributed to the degeneration and selective loss of dopaminergic neurons in the substantia nigra pars compacta (SNpc), leading to a dopamine (DA) deficiency in the striatum.

The environmental factors are the most common risk factor for Parkinson's disease, while hereditary determinants have minor role for disease. Furthermore, the clinical diagnosis of PD rests on the identification of characteristics related to dopamine deficiency. However, nondopaminergic and nonmotor symptoms, including cognitive dysfunction and depression, which is one of the most common and persistent symptoms, are sometimes present at an earlier disease stage and, almost inevitably, emerge with the disease progression.

Neuroinflammation is considered one of the most important factors contributing critically to pathophysiology of PD . Recently, high mobility group box-1 (HMGB1) protein has been encoded as a potential inflammatory biomarker in PD. HMGB1 mediates immune response mostly through endothelial cells and macrophage activation via targeting two vital cell receptors; Toll-like receptor 4 (TLR4) and advanced glycation end products (RAGE). HMGB1 leads to a sequential cascade of inflammatory response through enhanced release of tumor necrosis factor-alpha (TNF-α) and interleukins (ILs), prominently IL-1β and IL-6. HMGB1 mediated also up-regulation of nuclear factor kappa-β (NF-κB) with subsequent flared pro-inflammatory storm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both male and female will be included.
* Patients diagnosed with PD according to Unified Parkinson's Disease Rating Scale.

Exclusion Criteria:

* Breast feeding
* Patients with significant liver and kidney function abnormalities.
* Alcohol and / or drug abusers.
* Patients with known allergy to the study medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
- Change From Baseline for Unified Parkinson's Disease Rating Scale (UPDRS) Total Score | 6 months
  - Change From Baseline for Unified Parkinson's Disease Rating Scale (UPDRS) Total Score (Time Frame: Baseline and week 24)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Khrieba MO, Hegazy SK, Mohammed WF, El-Haggar SM. Clinical study to investigate the adjuvant role of Pentoxifylline in patients with Parkinson's disease: A randomized controlled study. Int Immunopharmacol. 2025 May 27;156:114689. doi: 10.1016/j.intimp.2025.114689. Epub 2025 Apr 19. PMID 40253769
- [Derived] Khrieba MO, Hegazy SK, Mustafa W, El-Haggar SM. Repurposing celecoxib as adjuvant therapy in patients with Parkinsonian disease: a new therapeutic dawn: randomized controlled pilot study. Inflammopharmacology. 2024 Dec;32(6):3729-3738. doi: 10.1007/s10787-024-01567-z. Epub 2024 Sep 28. PMID 39340691